CLINICAL TRIAL: NCT00394134
Title: A Targeted, Family-Focused Intervention for Melanoma Prevention
Brief Title: Targeted Intervention for Melanoma Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003-0901
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Melanoma
Keywords: Melanoma; Sun Exposure; Sun Protection; Interview
MeSH Terms: conditions — Melanoma | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Other): Interviews to describe the sun exposure and sun protection practices of patients and their children.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interviews to describe the sun exposure and sun protection practices of patients and their children.

SUMMARY:
In this study, the researchers will conduct interviews with melanoma patients to describe the sun exposure and sun protection practices of patients and their children. The researchers will use the findings of this interview study to develop a salient intervention targeted to the needs of melanoma patients and their children. The researchers will evaluate the intervention in a randomized, controlled trial.

The specific aims of this study are:

* To interview 210 melanoma patients with children 12 years of age or younger to describe patients' socio-cognitive and psychological factors, describe patients' and children's sun exposure and sun protection practices, and identify determinants of patients' and children's sun exposure and protective practices.
* To develop a targeted behavioral intervention that is designed to increase patients' protective practices to reduce their children's sun exposure, increase patients' self-protective practices, decrease the sun exposure levels of patients and their children, and positively influence socio-cognitive and psychological determinants of child-centered and self-protective practices.
* To conduct a randomized, controlled trial in a sample of 360 melanoma patients with children 12 years of age or younger to evaluate the targeted behavioral intervention consisting of print and video materials. The intervention will be assessed for its effects on: 1) child sun exposure and sun protection; 2) patients' protective practices to reduce their children's sun exposure; 3) patients' sun exposure and self-protective practices; and 4) patients' socio-cognitive and psychological factors that facilitate behavior change.

DETAILED DESCRIPTION:
Research is to learn about awareness, attitudes, and behaviors related to sun exposure, sun protection, skin examination, and other risk-reducing behaviors. The results of this study will be used to design an educational program on sun protection for persons who have had melanoma and their children.

The study will involve a telephone interview that will last about 45 minutes and will be scheduled at your convenience. Your participation in this study is completely voluntary and you may refuse to participate. Your decision about participating will not affect the care or services you or your family may receive at The University of Texas M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Melanoma patients are eligible if they were diagnosed with in situ, localized, or microscopic stage III melanoma after January 1, 1988.
2. Melanoma patients are eligible if they are the parent of a child 12 years of age or younger and reside with the child.
3. Melanoma patients are eligible if they provide informed consent.
4. Melanoma patients are eligible if they are 18 years of age or older.
5. Melanoma patients are eligible if they are able to speak, read, and write English.
6. Melanoma patients are eligible if they meet all inclusion criteria.

Exclusion Criteria:

1) Melanoma patients are not eligible if they cannot provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Patients'and Children's Sun Exposure and Protective Practices <Patient Interview Responses> | Baseline Interview, 6 Month and 9 Month Interviews
  Standard descriptive statistics computed for measures administered during structured interview, including means, standard deviations, ranges, measures of skew and kurtosis, together with 95% confidence intervals. Distributional characteristics of variables closely examined using boxplots, histograms, quantile-quantile plots, and the Kolmogorov-Smirnov test of normality.
  General linear mixed-model approach used evaluate associations between patient socio-cognitive factors, psychological factors, phenotypic characteristics, and demographic characteristics; child phenotypic and demographic characteristics; and practices of participants to reduce their children's sun exposure, self-protective practices of participants, and sun exposure practices of children and participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gritz ER, Tripp MK, Peterson SK, Prokhorov AV, Shete SS, Urbauer DL, Fellman BM, Lee JE, Gershenwald JE. Randomized controlled trial of a sun protection intervention for children of melanoma survivors. Cancer Epidemiol Biomarkers Prev. 2013 Oct;22(10):1813-24. doi: 10.1158/1055-9965.EPI-13-0249. PMID 24097199
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org